## Web-based Interpretation Training for Anxiety

## Informed Consent Form

NCT02382003

June 10, 2019

## IRB-SBS #2703 Consent

The purpose of this study is to investigate a new, experimental anxiety reduction program. It includes eight 20-minute sessions (some conditions will be faster, depending on your assignment), over the course of 3-4 weeks (2-3 sessions per week), and five 20-minute assessment sessions.

You will be presented with one of a few different training and/or imagery programs. We are testing which programs most effectively reduce anxiety. Although our prediction of which program will be most effective is based on previous work in the laboratory, we cannot be sure until the programs are compared by randomly assigning people to each one and then testing the effects. If you get randomly assigned to a program that we do not think will be the strongest one, you will then have the opportunity to complete the program we expect to be most effective after you finish the study. In other words, EVERYBODY gets a chance to try program we expect to be most effective eventually.

You will be asked to complete a 20-minute assessment before your 1st training session, after your 3<sup>rd</sup> training session, after your 6th training session, after your 8th training session, and 2 months after your 8th training session. The assessments will help us track your progress and determine if this new program is effective.

You will be asked to complete questionnaires in which you describe your thoughts and mood, describe your background and personal mental health history, and you may be asked to complete a task in which you read brief stories, answer questions, and complete word fragments. For some participants, being asked questions about their thoughts and mood can be temporarily distressing.

At the end of the study, you will receive more detail about the study's rationale and design. You will also receive feedback about the progress you made during the program and how your anxiety symptoms changed.

There may be no direct benefits to you. Depending on your randomly assigned condition, you may complete procedures that may help reduce symptoms of anxiety.

Remember that participation in this study is voluntary, and you may end your individual session participation at any time by closing the study window. Contact studyteam@mindtrails.org if you have any questions about the study, to withdraw completely from the study, or to receive payment after withdrawing.

Please note that MindTrails does not provide specific diagnostic or medical advice on our website, and we are limited in how we can respond to your personal requests .

Your responses will be confidential. We ask you to provide your email address and a user name (this can be your first name or any other name you choose), but your last name and mailing address are not required for this study.

Data collected through the MindTrails website are treated as confidential and are only accessible by the research team. The only exceptions to this guideline are if we learn of possible child abuse or neglect, or danger to self or others. In these instances,

confidentiality would be limited given mandated reporting requirements (e.g., to report the information to the police, or to child protective services).

## **Privacy Policy.**

MindTrails uses the same secure hypertext transfer protocol (HTTPS) that banks and other commercial websites use to transfer credit card information in an encrypted format. This provides strong security for data transfer to and from our website, though privacy is necessarily limited by the security of the technology that is being used. To view the entire privacy policy in a separate pop up window, please click here.

MindTrails is not able to offer financial compensation nor to absorb the costs of treatment should you feel you have been injured as a result of participating in the MindTrails research study.

To obtain more information about the study, ask questions about the research procedures, express concerns about your participation, or report illness, injury or other problems, please contact:

Tonya Moon, Chair, Institutional Review Board for the Social and Behavioral Sciences, One Morton Dr. Suite 500 University of Virginia, P.O. Box 800392, Charlottesville, VA 229080392. Telephone: (434) 924- 5999; Email: irbsbshelp@virginia.edu; Website: <a href="https://www.virginia.edu/vprgs/irb">www.virginia.edu/vprgs/irb</a>

By clicking the button below you are indicating that you have read the informed consent statement above and agree to participate.